CLINICAL TRIAL: NCT01162538
Title: The Main Objective of This Study is to Evaluate the Virologic Effectiveness at M6 of Regimen Containing Raltegravir in Treatment Naive HIV Subtype Non B or B Infected Subjects
Brief Title: To Evaluate Effectiveness and Safety of Containing Raltegravir in Naive HIV NON B or B Infected Patients
Acronym: Ral'inNONB
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Intercommunal Robert Ballanger (Other)
Responsible Party: Dr Jean-Luc Delassus, Réseau Aulnay 93
Other Study IDs: 2010-021178-12
Record Dates: First submitted 2010-07-09; First posted 2010-07-14 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-05

CONDITIONS: Evaluated; Non B Subtype; Naive Patients
Keywords: Raltegravir, non B subtype, naive patients

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Pilot open label multicentric study

DETAILED DESCRIPTION:
The population VIH1 not B is not unimportant in our region of the Seine St Denis, a tendency which seems to be in increase (47 % in 2006, 67 % in 2007).

Most of the studies evaluating the clinical, immunologic and virologic response to the ARV according to the viral subcategories are corresponding and show comparable results for patients infected by HIV 1 of subcategory B or non B. In spite of these reassuring results, it is necessary to evaluate the efficiency of a new ARV all the more a new class. It seems also necessary to observe attentively the profiles of resistance which will be selected at the carrier patient's of virus of subcategories not - B in failure of treatment. It will allow to determine if, because of the important polymorphisms of the viruses not - B, the evolution towards the resistance will be made differently.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to take part in this study, patients should meet all of the following criteria:

Patient aged at least 18 years; Treatment naive patient infected with HIV-1; Patients indicated for treatment containing raltegravir Patient has at least 2 activates molecules in combination therapy according genotype realized in the visit of selection.

Patient has not a history or current evidence of opportunist infection within the 4 weeks before the selection Patient who has received oral and written (information sheet) information about the study and who has agreed for the computer processing of his/her personal data.

Patients with chronic hepatitis, including chronic hepatitis B and/or C may enter the study as.

Exclusion Criteria:

* Patients meeting one or both of the following criteria may not take part in the study
* Patient is reproductive potential without requiring the use of contraception
* Patient is pregnant or breast-feeding
* Patient using alcohol and\or drug and\or the other substance that might interfere with the patient participation
* Patient infected by HIV2
* Patient has severe hepatic insufficiency. (liver enzymes > 5N)
* Patient has the following laboratory values during selection
* Platelets < 40.000 cell / mm3
* Haemoglobin < 8 g / dl during the selection
* Neutrophils < 500 / mm3
* Patient has associated treatments which can have interactions with Raltegravir (Cf RCP Isentress ®)
* Patient should be considered by the investigator able to conform to the imperatives of the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It's a pilot open label, multicentric, national, prospective and descriptive study to evaluate effectiveness and safety of regimen containing Raltegravir (400mg x 2) in 40 treatment naive HIV non B infected subjects versus in 20 treatment naive HIV B infected sujects.
  The patients will be matched according to:
  * basal viral load (< 10 000 copies/ml, ≥100 000 copies/ml)
  * rate of basal CD4 (<200 cell/mm3, ≥ 200 cell/mm3)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-03 (Estimated); Study Completion 2012-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Delassus Jean-Luc, MD, Principal Investigator — Réseau Aulnay 93
Locations (1):
- Hopital R.Ballanger, Aulnay-sous-Bois, France